CLINICAL TRIAL: NCT03230721
Title: Comparative Analysis of the Efficacy and Safety of Thulium-fiber Laser Enucleation, Ho:YAG Laser Enucleation and Monopolar Enucleation in Management of BPH
Brief Title: ThuLEP vs. HoLEP vs. Monopolar Enucleation in Management of BPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.M. Sechenov First Moscow State Medical University (Other)
Responsible Party: Principal Investigator, Dmitry Enikeev, MD, PhD, Deputy Director for Sсience, Dept. of Urology, I.M. Sechenov Moscow State Medical University, I.M. Sechenov First Moscow State Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMSechenovMMA
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Prostatic Hyperplasia, Benign; Prostate Adenoma; Lower Urinary Tract Symptoms
Keywords: laser; HoLEP; ThuLEP; Thulium; Thulium-fiber; BPH; EEP; monopolar enucleation
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ThuLEP group (Active Comparator): Patients who underwent thulium-fiber laser enucleation of the prostate due to lower urinary tract symptoms caused by prostatic hyperplasia.
  Interventions: Procedure: Thulium-fiber laser enucleation of the prostate
- Monopolar enucleation group (Active Comparator): Patients who underwent monopolar enucleation of the prostate due to lower urinary tract symptoms caused by prostatic hyperplasia.
  Interventions: Procedure: Monopolar enucleation of the prostate
- HoLEP group (Active Comparator): Patients who underwent Ho:YAG laser enucleation of the prostate due to lower urinary tract symptoms caused by prostatic hyperplasia.
  Interventions: Procedure: Ho:YAG laser enucleation of the prostate

INTERVENTIONS:
Procedure: Thulium-fiber laser enucleation of the prostate — A high-power (120 W) thulium fiber laser (Urolase, IPG IRE-POLUS, Russia) with wavelength of 1940 nm was used for thulium laser enucleation. In our study, we used a 600-μm laser fiber. The operations were performed at power of 60 W energy of 1.5 J and repetition rate of 40 Hz. Laser power in the verumontanum zone was decreased to 30 W and repetition rate to 20 Hz.
  Other Names: ThuLEP
  Arms: ThuLEP group
Procedure: Monopolar enucleation of the prostate — Monopolar enucleation was performed with a high-frequency generator (50-60 Hz), a pusher-electrode, and a hook-electrode.
  Other Names: Monopolar enucleation
  Arms: Monopolar enucleation group
Procedure: Ho:YAG laser enucleation of the prostate — Holmium laser enucleation of prostatic hyperplasia was performed with a 100 W laser (VersaPulse Powersuite 100, Lumenis, USA/Israel) with wavelength of 2100 nm and 550-μm fiber at the tip. The operation was performed at power of 70 W; it was decreased to 40 W when incisions were made at the verumontanum.
  Other Names: HoLEP
  Arms: HoLEP group

SUMMARY:
Today, endoscopic enucleation of the prostate (EEP) has been recognized a method of choice for treatment of benign prostatic hyperplasia (BPH) of any size, including large-sized glands (>80 cc). The goal of our study was to compare perioperative efficacy, functional outcomes and safety of different techniques of endoscopic enucleation of the prostate (monopolar enucleation, holmium laser enucleation, thulium laser enucleation) in a single center.

DETAILED DESCRIPTION:
HoLEP and ThuLEP or EEP have been approved by the current guidelines of the European Association of Urology for use in men with substantially enlarged prostates (>80 ml) as first-line therapy [1]. This type of operation can be performed by means of several sources of energy.

To our knowledge, there were no studies comparing efficacy and complications of these three treatment modalities.

In this study the investigators have evaluated efficacy of Thulium-fiber laser enucleation (120 W thulium fiber laser Urolase, IPG IRE-POLUS, Russia with wavelength of 1940 nm) and monopolar enuclation in comparision with HoLEP (VersaPulse Powersuite 100, Lumenis, USA/Israel) in reduction of LUTS secondary to BPH in a prospective randomized trial.

All peri-operative parameters, urinary flow parameters, prostate size changes, erectile function and complications associated with the procedures were compared.

ELIGIBILITY:
Inclusion Criteria:

* IPSS>20;
* maximum urinary flow rate< 10ml\s (Qmax);
* ineffective alfa-blockers therapy.

Exclusion Criteria:

* histologically verified prostate cancer;
* history of prostatic surgery;
* urethral strictures;
* bladder stones;
* chronic urinary retention and cystostomy.

Ages: 50 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 450 (Actual)
Dates: Start 2015-01-15 (Actual); Primary Completion 2017-04-22 (Actual); Study Completion 2017-07-21 (Actual)

PRIMARY OUTCOMES:
IPSS | Six months
  International Prostate Symptom Score

SECONDARY OUTCOMES:
QoL | Six months
  Quality of Life Score
PVR | Six months
  Post-void residual volume
Qmax | Six months
  Maximal urine flow rate
IIEF-5 | Six months
  The International Index of Erectile Function

CONTACTS AND LOCATIONS:
Overall Officials: Dmitry Enikeev, MD, PhD, Principal Investigator — I.M. Sechenov First Moscow State Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gratzke C, Bachmann A, Descazeaud A, Drake MJ, Madersbacher S, Mamoulakis C, Oelke M, Tikkinen KAO, Gravas S. EAU Guidelines on the Assessment of Non-neurogenic Male Lower Urinary Tract Symptoms including Benign Prostatic Obstruction. Eur Urol. 2015 Jun;67(6):1099-1109. doi: 10.1016/j.eururo.2014.12.038. Epub 2015 Jan 19. PMID 25613154
- [Background] Cornu JN, Ahyai S, Bachmann A, de la Rosette J, Gilling P, Gratzke C, McVary K, Novara G, Woo H, Madersbacher S. A Systematic Review and Meta-analysis of Functional Outcomes and Complications Following Transurethral Procedures for Lower Urinary Tract Symptoms Resulting from Benign Prostatic Obstruction: An Update. Eur Urol. 2015 Jun;67(6):1066-1096. doi: 10.1016/j.eururo.2014.06.017. Epub 2014 Jun 25. PMID 24972732
- [Background] Glybochko PV, Rapoport LM, Enikeev ME, Enikeev DV. Holmium laser enucleation of the prostate (HoLEP) for small, large and giant prostatic hyperplasia: tips and tricks. Urologia. 2017 Aug 1;84(3):169-173. doi: 10.5301/uj.5000232. Epub 2017 May 10. PMID 28497447